CLINICAL TRIAL: NCT01955902
Title: Using mHealth to Aid Opioid Medication Adherence Focus Groups
Brief Title: Using mHealth to Aid Opioid Addicts
Status: Completed | Type: Observational
Sponsor: Care Team Solutions (Industry)
Responsible Party: Sponsor
Other Study IDs: 271201300015C
Record Dates: First submitted 2013-09-26; First posted 2013-10-08 (Estimated); Last update posted 2013-11-11 (Estimated); Status verified 2013-11

CONDITIONS: Opiate Dependency Relapse
Keywords: Opioid dependence; Buprenorphine; Adherence; Substance use; Suboxone
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Opioid addicts: Opioid addicts undergoing bup/nal maintenance therapy

SUMMARY:
The purpose of the proposed study is perform focus groups to identify and prioritize features of the SubAID application (APP). The SubAID APP is smartphone APP being created to support patients self-managing buprenorphine/naloxone (bup/nal) medication. Many people have difficulty in managing bup/nal in the prescribed manner. Not taking medicines in their prescribed manner can cause negative health outcomes.

Focus group participants will be asked to elaborate on medication-taking patterns that work best for them, pitfalls associated with poor adherence and offer opinions upon what features/functions the SubAID APP should perform to be most helpful to them. The focus group is designed to remain open-ended and allow free discussion regarding each particular topic that the moderator will bring up.

DETAILED DESCRIPTION:
Opioid dependence (OD) is a serious medical and social quandary impacting the lives of millions, including disparate demographic populations in the United States. Economic and societal costs of prescription opioid abuse in the United States alone are estimated at $56 billion while the number of drug poisoning deaths attributed to opioid analgesics has more than tripled since 1999. In 2008, opioid analgesics were involved in greater than 40% of all drug poisoning fatalities. Opiate-agonist pharmacotherapy utilizing buprenorphine/naloxone (bup/nal) is known to decrease illicit opiate use. However, poor medication management and misuse during self-managed opioid substitution therapy (OST) constrains efficacy, while aggrandizing relapse, hospitalizations and mortality. In an adherence study, OST patients that mismanaged their medication were >10 times more likely to relapse than compliant patients. [5] Thus, one of the most inescapable challenges confronted by health care professionals treating OD is assuring medications are taken as prescribed to inhibit relapse. Yet, the threats to successful medication mismanagement for substance use disorders are unique from those of traditional chronic diseases.

While the ultimate goal of substance abuse treatment is abstinence, opioid addiction is a chronic, relapsing medical condition. Opioid substitution therapy, incorporating methadone or bup/nal, represents conventional treatment options for opioid dependence. Methadone maintenance in adequate doses reduces cravings, prevents the onset of withdrawal, is not intoxicating or sedating, and does not interfere with normal activities of daily living. However, significant pitfalls denote methadone maintenance treatment. Methadone is a long-acting, full opioid agonist with known abuse and diversion potential and no upper boundary to the level of respiratory depression -- overdose can therefore be fatal. In addition, relapse rates for methadone maintenance range between 55-90% following treatment. Although an effective therapy, the high rates of relapse and diversion render methadone a less than ideal solution for many patients. Recently, the bup/nal formulation, commonly sold as Suboxone®, was designed to minimize abuse and diversion while retaining all positive aspects of methadone treatment. Bup/nal has proven correspondingly effective in treating OD as methadone, and more efficient in certain populations. Clinical studies have shown the beneficial effect of bup/nal treatment in reducing subsequent opioid use. Administered sublingually, naloxone undergoes extensive first-pass metabolism and has negligible bioavailability; thus, when used as prescribed, the combination drug (bup/nal) produces effects of buprenorphine alone. However, if injected, the naloxone will precipitate withdrawal in opioid dependent patients. Thus, bup/nal is intended to reduce the risk of illicit use by injection. An additional benefit of bup/nal OST is unsupervised use. Unlike methadone maintenance, which generally entails a daily clinic visit, bup/nal allows the patient increased freedom, typically requiring only one physician and pharmacy visit per month after a stabilization period. Given its lower abuse appeal, strong effectiveness, and clear ability to lower relapse rates, bup/nal represents a more suitable treatment option for OD, especially in still working individuals.

In spite of moves toward more unsupervised and self-managed OST with bup/nal, monitoring and promoting effective medication adherence is challenging for a number of reasons including diversion, lack of motivational support to avoid opioids, and low health literacy. Affording patients and their caregivers an interactive toolset to effectively monitor and promote medication management during OST therefore represents a major unmet need that this project will address. This research project will develop an interactive smartphone/tablet application (APP), named SubAID, designed to engage and support patients receiving bup/nal to promote and monitor adherence. In order to develop the most appropriate and effective adherence support content for the SubAID APP, we will solicit opinions in Focus Groups from OD subjects prescribed bup/nal to better understand the adherence complications and problems they encounter on a daily basis.

ELIGIBILITY:
Inclusion Criteria:

* At least 21 years of age
* Physician diagnosis of opioid dependence (OD)
* Prescribed buprenorphine/naloxone (bup/nal) and acclimated to the medication
* Able to speak and read English
* Willing to provide written informed consent prior to study entry
* Able to understand the study
* Ownership of an Android or iPhone smartphone

Exclusion Criteria:

* Having any concurrent medical or psychiatric condition that, in the investigator's opinion, may preclude participation in this study; or
* Cognitive or other impairment (e.g., visual) that would interfere with completing a self-administered questionnaire and with participating in a group discussion.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community Sample
Sampling Method: Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2013-08; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Attitudes, beliefs and perceptions | Up to 8 weeks
  Content analysis will be used to evaluate the information gathered during the focus groups. The analysis will be based on recall, notes taken by the co-facilitator, and transcripts from session recordings. The evaluation process will include the following: 1) generation of key words, phrases, and quotes concerning symptoms, concerns or fears about their ability to effectively manage maintenance medications, and 2) identification of additional, emergent themes in each of the SubAID features that would be helpful and relevant to the impact of managing maintenance therapy medications. To be considered credible, themes included in the final analysis will be features or concerns that were raised by more than one participant in a single group, and, ideally, by participants in more than one group.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bailey, PhD, Study Director — Care Team Solutions
Locations (1):
- Care Team Solutions, Lexington, Kentucky, United States